CLINICAL TRIAL: NCT03843424
Title: A Pragmatic Family-Centered Approach to Childhood Obesity Treatment
Brief Title: Treatment Efforts Addressing Child Weight Management by Unifying Patients, Parents & Providers
Acronym: TEAM UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Blue Cross and Blue Shield of Louisiana (Unknown); American Academy of Pediatrics (Other); Pennington Biomedical Research Center (Other); Louisiana Healthcare Connections (Unknown); Nationwide Children s Hospital in Columbus, Ohio (Unknown); University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201810158; PCS-2017C2-7542 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Obesity, Childhood; Pediatric Obesity; Childhood Obesity; Adolescent Obesity; Overweight; Overweight and Obesity; Overweight or Obesity; Overweight Adolescents; Weight Gain; Overnutrition; Body Weight; Body Weight Changes; Nutrition Disorders
Keywords: Weight Management; Child; Intervention; Weight Loss; Behavior Therapy; Nutrition
MeSH Terms: conditions — Pediatric Obesity; Overweight; Obesity; Weight Gain; Overnutrition; Body Weight; Body Weight Changes; Nutrition Disorders; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Standard of Care (eSOC) (Active Comparator): This group will receive the eSOC program. A minimum of 6 visits to the primary care provider (PCP) and includes assessment of weight status, patient/family motivation and readiness to change, promotion of healthy eating and activity habits, and use of health behavior change strategies.
  Interventions: Behavioral: eSOC program
- Family-Based Behavioral Treatment (FBT + eSOC) (Active Comparator): This group will receive eSOC plus the FBT program. Family-based behavioral treatment (FBT), an effective treatment that targets both child and parents meeting regularly with a health coach for healthy eating, activity, positive parenting strategies, and managing environmental cues.
  Interventions: Behavioral: eSOC program; Behavioral: FBT program

INTERVENTIONS:
Behavioral: eSOC program — American Medical Association (AMA) recommended staged approach to childhood obesity screening and counseling
Behavioral: FBT program — An intensive,comprehensive, behavioral intervention aligned with the US Preventive Services Task Force recommendations for childhood obesity screening and counseling.
  Arms: Family-Based Behavioral Treatment (FBT + eSOC)

SUMMARY:
The US Preventive Services Task Force (USPSTF) recommends that providers screen children aged 6 years and older for obesity and offer or refer them to a comprehensive behavioral intervention (≥26 hours over a period of up to 12 months) to promote improvement in weight status. Family-based behavioral treatment (FBT) is an effective treatment that targets both child and parents and meets the USPSTF recommendations. By contrast, the American Medical Association (AMA) recommends a staged approach to childhood obesity screening and counseling, which begins with prevention counseling by the primary care provider (PCP) and includes assessment of weight status, patient/family motivation and readiness to change, promotion of healthy eating and activity habits, and use of health behavior change strategies. Our study compares a staged approach enhanced standard of care (eSOC) vs. eSOC + FBT, to provide families and PCPs with information on the best intervention approach for the behavioral treatment of childhood obesity. Our project seeks to fill the gap in the evidence on family-based weight management in primary care settings among diverse and underserved populations with a special focus on Black children, families insured by Medicaid, and sex differences.

DETAILED DESCRIPTION:
Note: our enrollment number includes two participants (one child and one parent) from each enrolled family.

ELIGIBILITY:
Inclusion Criteria for children include:

* have a BMI percentile ≥95th for age and sex;
* comfortable speaking English language;
* able to provide written or verbal (based on age) informed assent;
* willing to change diet, physical activity, and/or weight;
* patient of a participating clinic/practice; and
* able to participate in scheduled sessions.

Inclusion Criteria for parents include:

• comfortable speaking and reading English language.

Exclusion Criteria include:

* families who plan to no longer have the child be a patient of any participating clinic/practice during any point in the 18-month study period;
* children with chronic conditions or on medications that substantially impact or interfere with growth, appetite, weight, or physical activity participation;
* families for whom the Primary Care Provider (PCP) or site PI thinks the intervention is clinically/medically inappropriate (e.g., developmental delay, or emotional or cognitive difficulties, if the PI/PCP believes these factors will interfere with study/intervention participation); and
* families in whom the parent or child exhibits eating disorder symptomatology.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1460 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Child percent overweight | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Denise E. Wilfley, PhD, Principal Investigator — Washington University School of Medicine; Stephen Cook, MD, MPH, Principal Investigator — University of Rochester
Locations (7):
- United States (7):
  - Washington University School of Medicine, Alton, Illinois
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Pennington Biomedical Research Center, New Orleans, Louisiana
  - Washington University School of Medicine, Cape Girardeau, Missouri
  - University of Missouri School of Medicine, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York

REFERENCES:
- [Derived] Staiano AE, Button AM, Baker A, Beyl R, Conn AM, Lima A, Lindros J, Newton RL Jr, Stein RI, Welch RR, Cook S, Wilfley DE; TEAM UP Research Group. A pragmatic trial of a family-centered approach to childhood obesity treatment: Rationale and study design. Contemp Clin Trials. 2024 Mar;138:107459. doi: 10.1016/j.cct.2024.107459. Epub 2024 Jan 24. PMID 38278478